CLINICAL TRIAL: NCT06732362
Title: To Observe the Clinical Effect of Femoral Nerve Block With Low Concentration Ropivacaine Under Ultrasound Guidance Combined With Neurostimulator Based on DPN Grading
Brief Title: To Observe the Clinical Effect of Femoral Nerve Block With Low Concentration of Ropivacaine Based on DPN Grading
Status: Not yet recruiting | Type: Observational
Sponsor: Zheng Guo (Other)
Responsible Party: Sponsor-Investigator, Zheng Guo, Chief physician, Second Hospital of Shanxi Medical University
Organization: Second Hospital of Shanxi Medical University (Other)
Other Study IDs: HanYi20241211
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- No peripheral vascular neuropathy: Grouping was performed according to the TCSS grading scale
  Interventions: Other: Different DPN ratings
- Mild peripheral vascular neuropathy: Grouping was performed according to the TCSS grading scale
  Interventions: Other: Different DPN ratings
- Severe peripheral vascular neuropathy: Grouping was performed according to the TCSS grading scale
  Interventions: Other: Different DPN ratings

INTERVENTIONS:
Other: Different DPN ratings — According to the TCSS grading scale, DPN patients were graded into different grades, and the mild and severe groups and the control group were selected to observe the clinical effects between the three groups

SUMMARY:
The purpose of this study was to quantitatively standardize the performance of patients with DPN with different course of disease using high-frequency ultrasound, and to design experiments to verify the conclusion that DPN patients with peripheral nerve damage increased nerve sensitivity to local anesthetic drugs and increased block time, and to achieve the same blocking effect by using low-concentration local anesthetic drugs, so as to reduce the probability of complications such as transient nerve injury, severe nerve injury, and local anesthetic poisoning.

DETAILED DESCRIPTION:
Clinically, through the correlation study between the serum choliphin concentration and the degree of neuropathy (cross-sectional area) of patients with DPN (scale standardization) of different course of disease and the degree of neuropathy under ultrasound, the DPN was standardized after conclusion, and then the clinical study was designed to use low concentrations of ropivacaine to perform nerve blocks at the same site in patients with DPN of different grades, and the time t of the first use of the analgesic pump after the primary outcome measures, the electrical stimulation threshold during nerve block, and the secondary outcome indicators were the threshold of electrical stimulation during nerve block, Sensory and motor block time-to-occur to assess the effect of nerve block.

ELIGIBILITY:
Inclusion Criteria:All patients met the 1999 WHO diagnostic criteria for diabetes.

-

Exclusion Criteria:(1) Type 1 diabetes; (2) Peripheral neuropathy obviously caused by other reasons; (3) Patients with neuropathy caused by diabetic foot ulcers and gangrene, as well as known history of bone and joint trauma or surgery of the lower limbs; (4) Contraindications to peripheral nerve block (such as local anesthetic allergy, coagulation dysfunction, peripheral infection, etc.) (5) Contraindications to drug components of postoperative analgesic pumps; (6) Existing opioid therapy.

-

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in the Second Hospital of Shanxi Medical University from December 2024 to June 2025
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-10-29 (Estimated)

PRIMARY OUTCOMES:
N/OFQ | 24 hours
  Serum N/OFQ levels

SECONDARY OUTCOMES:
Time to onset of nerve block | 24 hours
  The sensorimotor disappearance time was observed after self-administration
Ratio of femoral nerve to femoral artery cross-sectional area | 24 hours
  The ratio of the two was measured to observe the change

CONTACTS AND LOCATIONS:
Overall Officials: yi Han, Doctor, Study Director — Second Hospital of Shanxi Medical University
Locations (1):
- Second Hospital of Shanxi Medical University, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No